CLINICAL TRIAL: NCT02651025
Title: Effects of Resistance Training on Physical Activity in Daily Life, Muscle Function and Functional Capacity in Patients With End Stage Renal Disease on Hemodialysis: a Randomised Controlled Trial
Brief Title: Effects of Resistance Training on Physical Activity in Daily Life and Functional Capacity in Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Juiz de Fora (Other)
Responsible Party: Principal Investigator, Maycon de Moura Reboredo, Professor of School of Medicine, Federal University of Juiz de Fora
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE:44426115.0.0000.5147
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistance Exercise Program (Experimental): Patients included in intervention group will submit to resistance exercise training during hemodialysis, three times a week, for twelve weeks. This program includes exercises for the upper and lower limbs.
  Interventions: Other: Resistance Exercise Program
- Passive Stretching Program (No Intervention): Patients included in control group will submit to passive stretching program of lower limbs, during hemodialysis, three times a week, for twelve weeks.

INTERVENTIONS:
Other: Resistance Exercise Program — During the first week of training will be conducted two sets of 10 repetitions, and from the second week of training until the twelfth will be performed three sets of 10 repetitions. The work rate will set to the tolerance of each patient as established by his/her inability to maintain Borg ratings for dyspnea and effort (10-point category-ratio Borg scale) scores between "4" and "6".
  Arms: Resistance Exercise Program

SUMMARY:
The purpose of this study is to determine whether a supervised resistance exercise training during hemodialysis is effective to increase physical activity in daily life in patients with end stage renal disease.

DETAILED DESCRIPTION:
The patients will be randomized into two groups: intervention and control groups. Patients in the intervention group will receive a supervised resistance exercise training, during hemodialysis, three times/week for 12 weeks, and patients allocate to the control group will received a passive stretching program during the same timeframe.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end stage renal disease on hemodialysis for at least three months
* Sedentary for at least six months

Exclusion Criteria:

* Presence of physical limitations that prevent the implementation of physical tests
* Presence of severe comorbidity and unstable (unstable angina, decompensated heart failure, myocardial infarction history of the past six months, cardiac arrhythmias, uncontrolled hypertension with systolic blood pressure ≥ 200 mmHg and / or diastolic blood pressure ≥ 120 mmHg, diabetes decompensated, severe lung disease, acute systemic infection as well as neurological disorders, musculoskeletal and osteoarticular or other disabling conditions according to the clinical judgment)
* Hospitalization in the three months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Physical Activity in Daily Life | 12 weeks
  The physical activity in daily life will be estimated as the mean number of steps using a triaxial accelerometer.

SECONDARY OUTCOMES:
Muscle function | 12 weeks
  The muscle function will be assessed by electromyography.
Muscle strength | 12 weeks
  The measurement of maximal voluntary strength of handgrip will be assessed by hydraulic model of dynamometer.
Functional capacity | 12 weeks
  The functional capacity will be assessed by six-minute walking test.
Quality of life | 12 weeks
  The quality of life will be assessed by the 36-Item Short Form Health Survey (SF36).
Depression and anxiety | 12 weeks
  Depression and anxiety will be assessed by the Hospital Anxiety and Depression Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Maycon M Reboredo, DSc, Study Director — Federal University of Juiz de Fora; Felipe M Valle, Principal Investigator — Federal University of Juiz de Fora; Bruno V Pinheiro, DSc, Study Director — Federal University of Juiz de Fora
Locations (1):
- University Hospital of the Federal University of Juiz de Fora, Juiz de Fora, Minas Gerais, Brazil

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639